CLINICAL TRIAL: NCT06115317
Title: Homonymous Hemianopia in Childhood
Acronym: HHIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 18BA25
Record Dates: First submitted 2023-08-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Homonymous Hemianopia
Keywords: Homonymous Hemianopia; Children and Young People
MeSH Terms: conditions — Hemianopsia | interventions — PRDM6, protein, mouse; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Double blind cross over.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prism followed by sham (Other)
  Interventions: Other: Prism; Other: Sham
- Sham followed by prism (Other)
  Interventions: Other: Prism; Other: Sham

INTERVENTIONS:
Other: Prism — Prism
Other: Sham — Sham

SUMMARY:
The study will consist of two connected components at a single centre. Phase 1 is observational, phenotyping children with Homonymous hemianopia (HH). Phase 2 is a pilot double blind cross over RCT in which segmental prisms are compared with sham prisms in glasses.

DETAILED DESCRIPTION:
The project will consist of two connected pieces of work. The primary phase of the study will examine children with a diagnosis of homonymous hemianopia to investigate the clinical spectrum, and undertake questionnaires to measure vision related quality of life and visual function. Functional evaluation will also include optical coherence tomography, electrophysiological and eye movement studies.

If the recruited children or young people meet the inclusion criteria for phase two they will then be given the option of taking part in phase 2 - a pilot randomised cross-over trial of prism glasses. The order in which the prism lenses and the sham lenses are given will be randomised, with each worn for four weeks. The child or young person and their parent carer will be asked for their opinion on each pair, with the primary outcome question "If the trial was to end today would you want to continue wearing these lenses?" (Yes/no). Visual function will be measured behaviourally using a questionnaire based tool, and functionally utilising an eye movement recording of a visual search task.

The project consists of two connected studies. The primary phase of the study will examine children with homonymous hemianopia to investigate the spectrum of eye features. This will involve doing several different eye tests, similar to ones used in clinical practice. All children will have a photo of their eye taken that measures the thickness of the nerve at the back of the eye. They will also have electrodes put on their head and around their eyes that will measure the brains response to different visual stimuli. This is not painful and they children can choose a carton to watch during it to make it more entertaining. The children will also have their eye movements measured as they follow a target on a TV screen towards the non-seeing and seeing half of the vision. The children will also be asked to do some drawing tasks such as putting numbers on a clock face, or drawing a house to see how much they do or don't ignore the side with the visual impairment. They will also undertake age appropriate questionnaires to measure their vision related quality of life and visual function. This will give us more information about what impact the HH has on different aspects of their lives.

If the recruited children in phase 1 meet the inclusion criteria for phase 2 they will be invited to take part. Phase 2 is a trial of prisms glasses. Participants will be told they are trialing two different pairs of glasses one with the full prism and one with a weaker (sham) prism, and will be unaware which one is which, as will the study investigator. The order in which they wear the glasses will be random. They will wear each pair for four weeks and return for an assessment at the end of each four weeks of wear. At each assessment the children will complete a questionnaire to measure if or how the glasses helped them.

They will also have their eye movements measured to see if they make more compensatory movements towards the blind side. Patient's opinions will also be recorded including responses to the question "If the trial was to end today would you want to continue wearing these glasses?".

ELIGIBILITY:
Inclusion Criteria:

Phase 1 inclusion criteria:

1. Clinical diagnosis of homonymous hemianopia
2. Age 5 to 17
3. Corrected visual acuity within normal limits for age,
4. No evidence of eye pathology (pathology of the eye its self that causes additional visual impairment on top of the homonymous hemianopia) including no nystagmus
5. No marked refractive error > +/-5.00DS
6. Complete homonymous hemianopia of more than 6 months - to avoid any natural recovery or adaptation (i.e. in stroke)

Phase 2 inclusion criteria:

1. Participation in phase 1 or copy of a detailed clinical assessment in the last 6 months from GOSH or a PIC site.
2. No hemispatial visual neglect detected in phase one or a clinical assessment
3. Aged 7 to 17
4. Corrected visual acuity within normal limits for age,
5. No evidence of eye pathology (pathology of the eye its self that causes additional visual impairment on top of the homonymous hemianopia) including no nystagmus
6. No marked refractive error > +/-5.00DS
7. Complete homonymous hemianopia of more than 6 months - to avoid any natural recovery or adaptation (i.e. in stroke)

Exclusion Criteria:

Phase 1 exclusion criteria:

1. Cannot establish definite clinical diagnosis of homonymous hemianopia
2. Have participated in other studies undertaking intervention for homonymous hemianopia
3. Reduced corrected visual acuity for age and/or high glasses prescription.
4. Eye pathology (that causes additional visual impairment to the homonymous hemianopia) and/or nystagmus
5. Homonymous hemianopia incomplete or less than 6 months old
6. Suspected or proven deficit of the unaffected hemisphere of the brain

Phase 2 exclusion criteria:

1. No participation in phase 1 or copy of a detailed ophthalmology assessment in the last 6 months from GOSH or a PIC site.
2. Hemispatial visual neglect
3. Cannot establish definite clinical diagnosis of homonymous hemianopia
4. Age/ability/additional disability means cannot give subjective responses
5. Have participated in other studies doing intervention for homonymous hemianopia
6. Reduced corrected visual acuity for age and/or high glasses prescription
7. Eye pathology (that causes additional visual impairment to the homonymous hemianopia) and/or nystagmus
8. Homonymous hemianopia incomplete or less than 6 months old
9. Suspected or proven deficit of the unaffected hemisphere of the brain

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Is it possible to run a full randomised control trial of the use of segmental prisms in children with Homonymous Hemianopia? | 2 years
  My primary outcome is asking participants "if the trial ended would you want to continue wearing these glasses?"

SECONDARY OUTCOMES:
Is it possible to run a full randomised control trial of the use of segmental prisms in children with Homonymous Hemianopia? | 2 years
  Recruitment rates using descriptive statistics.
Is it possible to run a full randomised control trial of the use of segmental prisms in children with Homonymous Hemianopia? | 2 years
  Retention rate using descriptive statistics.
Is it possible to run a full randomised control trial of the use of segmental prisms in children with Homonymous Hemianopia? | 2 years
  Reporting any harms or unintended effects (descriptive statistics).

CONTACTS AND LOCATIONS:
Overall Officials: Jugnoo Rahi, Principal Investigator — GOSH Institute of Child Health
Locations (1):
- Great Ormond Street Hospital for Chidlren, London, United Kingdom